CLINICAL TRIAL: NCT00832325
Title: Adolescent and Young Adult Cancer Survivors: Identity Development
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09-001
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Childhood Survivor; survivors; Young Adult Cancer Survivors; Childhood cancers; 09-001
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic; Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- 1 individual interviews: The patient will be asked to come in to the Counseling Center at MSKCC (641 Lexington Avenue, 7th Floor) and participate in an individual interview at their convenience.
  Interventions: Behavioral: interview
- 2 Focus Groups: The patient will be asked to come in to the Counseling Center at MSKCC (641 Lexington Avenue, 7th Floor) and participate in a focus group at their convenience.
  Interventions: Behavioral: Focus groups
- 3 Questionnaire: The patient will be asked to participate in three 60-90 minute telephone interviews scheduled at their convenience.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: interview — The doctor and/or one of her trained research study staff will ask the patient about their experience as an adolescent/young adult cancer survivor, their health and quality of life. It should take (approximately 1-1 ½ hours)to complete. Interviews will be audiotaped and transcribed by a professional transcription service.
  Groups: 1 individual interviews
Behavioral: Focus groups — The patient will participate with 6-8 other adolescent/young adult cancer survivors. The doctor and/or her trained research study staff will ask about their experience as an adolescent/young adult cancer survivor, their health and quality of life. It should take about one-and-a-half hour to complete. Focus groups will be audio taped and transcribed by a professional transcription service.
  Groups: 2 Focus Groups
Behavioral: Questionnaire — The patient will be asked to participate in three 60-90 minute telephone interviews conducted by the doctor and/or her trained research study staff scheduled at the patient's convenience, the second interview approximately 6-8 months after the first and the last interview approximately 12-16 months after the first. The questionnaire will ask about their experience as an adolescent/young adult cancer survivor, their health and quality of life.
  Groups: 3 Questionnaire

SUMMARY:
The purpose of this study is to better understand how the illness has affected the identity and what needs the survivor may have. We hope that this information will help us provide better care to future adolescent and young adult cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Current age greater than and including 15 and up to and including 25 years of age at time of consent
* Diagnosis of a first cancer > or = to 14 and up to and including 21 years of age
* At least 6 months post-treatment according to participant's self-report.
* Able to provide informed consent (or parent or legal guardian consent and participant assent for those participants under 18 years of age)
* Able to speak English. This inclusion criterion is included because study assessments were designed and validated in English and many of them are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the assessments.

Exclusion Criteria:

* Will exclude survivors with severe cognitive impairment that precludes them from being able to give information consent and/or complete the questionnaires.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: adolescent survivors from MSKCC
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-01; Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Conduct a comprehensive qualitative assessment through individual interviews and focus groups of identity development, peer and family relationships, and psychosocial concerns among survivors diagnosed during adolescence. | 3 years

SECONDARY OUTCOMES:
Conduct a prospective longitudinal assessment of identity development and peer and family relationships among survivors diagnosed during adolescence. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Marie Barnett, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org